CLINICAL TRIAL: NCT00708240
Title: Treatment With Escitalopram (Cipralex®) for Adolescents With Obsessive-Compulsive Disorder: Efficacy, Safety, and Changes in Executive Functions, Metacognition, and Regional Brain Activations.
Brief Title: Treatment Youth With Obsessive-Compulsive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Martine F. Flament, Univeristy of Ottawa Institute of Mental Health Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMHR-REB-2006-14
Record Dates: First submitted 2008-06-26; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escitalopram (Experimental)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram will be provided in unit doses commercially available, with a starting dose, minimum effective dose, and maximum effective dose of 5 mg, 10 mg and 20 mg, respectively, given once daily.
  Other Names: Cipralex

SUMMARY:
Although research suggests that patients with obsessive-compulsive disorder (OCD) exhibit specific deficits in their high cognitive processes, it is still unknown how these deficits relate to the clinical symptoms of the disorder, and to the response to treatment. There are two aims for the proposed research. The first is to examine how high cognitive processes and brain activity are affected in OCD. The second aim is to investigate the effects of a specific psychotropic medication (escitalopram) on high cognitive processes and brain activity in OCD. We will investigate how 40 youth with OCD (recruited in specialized clinics) differ from 40 healthy youth (recruited from the local community) on selected cognitive tests and brain imaging paradigms, as well as explore how treatment with medication can correct or reverse the observed differences. The final goal of our research is to learn more about the mechanisms of action for available treatments, in order to refine and improve short- and long-term therapeutic strategies for a highly debilitating and often lifelong disorder.

DETAILED DESCRIPTION:
Rationale. Obsessive-compulsive disorder (OCD) often has a childhood onset, and is characterized by recurrent obsessions and compulsions that are perceived as irrational and cause significant interference in daily functioning. Neuropsychological and/or neuroimaging investigations have consistently implicated pathways involving the ventral prefrontal cortical regions in the pathophysiology of the disorder. In the absence of attention or memory loss, OCD patients perform more poorly than controls on tasks requiring inhibition of an automatic response. Dysfunction of a frontal-striatal-thalamic circuit in OCD may be mediated by abnormalities in glutamatergic-serotonin neurotransmission, and selective serotonin reuptake inhibitors (SSRIs) are the unique class of psychotropic medication with demonstrated efficacy for youth (and adults) with the disorder.

Objectives and hypotheses. The first objective of the study is to examine how executive functions, metacognition performance, and regional brain activations differ in adolescents with OCD compared to healthy controls. Three specific hypotheses will be tested: (1) in adolescents with OCD, the executive functions related to the frontal cortex will be impaired compared to healthy controls; (2) the metacognition performance of the OCD group will be lower than that of the control group; (3) using fMRI, the OCD group's frontal lobe activations during tasks testing response inhibition and working memory, will be higher than those in the control group. The second objective is to investigate how treatment with the SSRI escitalopram will affect executive functions, metacognition performance, and regional brain activations in adolescents with OCD. After pharmacotherapy, three specific hypotheses will be tested: (1) there will be significant improvement from baseline in the OCD group's frontal executive functions and metacognition performance; (2) the differences on executive functions and metacognition performance between the OCD and control groups will no longer be significant; (3) on repeated fMRI procedures, the OCD group's frontal lobe activations will show a significant decrease from baseline. The third objective is to explore, within the patient group, the relationships between the degree of clinical change, and the magnitude of pre-post-treatment changes in neurocognitive performance, and regional brain activations. The hypothesis is that greater clinical improvement will be associated with greater changes on the selected neurocognitive and neurofunctional measures.

Method. Forty subjects, aged 13-19 years, with a primary DSM-IV diagnosis of OCD, and 40 sex-, and age-matched healthy controls, will be recruited from Ottawa mental health centers and the community. The study will use a pre- post-treatment design, and include three phases. Phase I: Pre-treatment, the OCD subjects will be compared to controls on clinical, neurocognitive, and functional brain activation measures. Phase II: The OCD subjects will receive open treatment with escitalopram (5 mg to 20 mg/day) for 16 weeks. Phase III: The clinical, neurocognitive, and functional brain activations measures will be repeated in all OCD subjects who completed 16 weeks of escitalopram pharmacotherapy, and the neurocognitive measures in control participants after 16 weeks. The Wisconsin Card Sorting Test, Stroop Test, and a Working Memory Task will be used to assess frontal executive functions. The Feeling-of-knowing task and Metacognition Questionnaire will measure metacognition performances. To investigate regional brain activations (only in participants aged 15-19 years), two functional neuroimaging paradigms will be used, a Go/NoGo and a n-Back task, and regional brain activations will be measured using fMRI technology. In patients, clinical severity and changes with treatment will be assessed using the Children's Yale Brown Obsessive-Compulsive Scale, the Maudsley Obsessive-Compulsive Inventory, the State-Trait Anxiety Inventory for Children, and the Children Depression Inventory. Statistical methods will include repeated measures MANOVAS, t-tests, and correlational analyses.

ELIGIBILITY:
Inclusion Criteria:

* Be 13 to 19 years old
* Have at least average intellectual ability
* Currently meet DSM-IV-TR criteria for OCD, upon completion of the Anxiety Disorder Interview Schedule for DSM-IV - Research and Lifetime Version for child and parent (ADIS- RLV)
* Receive a total score equal to or greater than 20 on the CY-BOCS at the screening visit have less than 25% decrease on the CY-BOCS total score between the screening and baseline visit
* If female of childbearing potential and sexually active in a heterosexual relationship, the subject must be using a reliable method of contraception, such as hormonal contraceptives
* Oral contraceptives must have been started at least 3 months prior to the start of the study

Exclusion Criteria:

* Clinically significant and/or unstable medical condition, including cardiovascular, respiratory, hematological, neurological and endocrine diseases
* History of neurological disorder or head injury
* Current use of medication with central nervous system effects
* Substance abuse or dependence within 6 months prior to enrolment
* Contra-indication to the fMRI
* Color blindness
* A comorbid current DSM-IV Axis I diagnosis, except for tic disorders and another anxiety disorder, as long as the associated disorder is less disabling than the primary diagnosis of OCD, as can be assessed with the ADIS
* Patients who would require additional psychological or pharmacological treatment
* Significant suicide risk, based on clinical judgment and the relevant section of the ADIS
* Hypersensitivity to escitalopram
* Previous non-response to an adequate trial of escitalopram
* Any lifetime psychiatric disorder as assessed on the ADIS
* A lifetime diagnosis of schizophrenia in biological parents or siblings

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-08 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale score. | Before and after treatment and at each study visit

SECONDARY OUTCOMES:
Clinical Global Impression for Severity of Illness and Improvement | each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Martine F. Flament, MD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa Institute of Mental Health Research, Ottawa, Ontario, Canada